CLINICAL TRIAL: NCT04682626
Title: Effect of Weekly High-dose Vitamin D3 Supplementation on the Association Between Circulatory FGF-23 and A1c Levels in People With Vitamin D Deficiency
Brief Title: Effect of Weekly High-dose Vitamin D3 Supplementation on the Association Between Circulatory FGF-23 and A1c Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Principal Investigator, Mahmoud Suleiman Abu-Samak, Mahmoud S Abu-Samak, PhD Study Principal Investigator Department of Clinical Pharmacy and Therapeutics, Applied Science Private University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-PHA-23
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2; Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VD3 group (Experimental): Dietary Supplement: Soft gelatin capsules each contain 50 000 IU VD3 (cholecalciferol) equivalents to 1.25 mg once weekly for 8 weeks.
  .
  Interventions: Dietary Supplement: Soft gelatin capsules each contains 50 000 IU VD3 (cholecalciferol) equivalents to 1.25 mg.
- Control group (No Intervention): none has been administered

INTERVENTIONS:
Dietary Supplement: Soft gelatin capsules each contains 50 000 IU VD3 (cholecalciferol) equivalents to 1.25 mg. — Soft gelatin capsules each contain 50 000 IU VD3 (cholecalciferol) equivalents to 1.25 mg.
  Arms: VD3 group

SUMMARY:
Among Jordanians, there is a high prevalence of T2DM. VDD has also spread rapidly in the past decade. Preliminary results of recent studies have shown that VD3 has a potential role in reducing FBG. Notably, the impact of VD3 supplementation on glycemic control in diabetics, as well as pre-diabetics, remains highly controversial. Some studies have shown that osteocalcin (OSC) is correlated with fat mass, sensitivity to and secretion of insulin, glucose metabolism, and glycemic variability. In mice, OSC injections improved insulin sensitivity and prevent obesity. A more recent study has found that T2DM was inversely correlated with osteocalcin levels . There is a strong correlation between OSC and fibroblastic factor -23 (FBF-23). Many recent studies have correlated FBF-23 as well as vitamin D levels with some of the pathological conditions such as chronic kidney failure, atherosclerosis, and diabetes. They stated possible interrelationships between insulin resistance, Hyperinsulinemia, and/or lower VD3 levels may lead to decreased serum FGF-23 concentrations in obese children and adolescents. Therefore, serum FGF-23 has been suggested to be a potential indicator of subclinical atherosclerosis in patients with gestational diabetes mellitus.

DETAILED DESCRIPTION:
Among Jordanians, there is a high prevalence of T2DM. VDD has also spread rapidly in the past decade. Preliminary results of recent studies have shown that VD3 has a potential role in reducing FBG. Notably, the impact of VD3 supplementation on glycemic control in diabetics, as well as pre-diabetics, remains highly controversial. Some studies have shown that osteocalcin (OSC) is correlated with fat mass, sensitivity to and secretion of insulin, glucose metabolism, and glycemic variability. In mice, OSC injections improved insulin sensitivity and prevent obesity. A more recent study has found that T2DM was inversely correlated with osteocalcin levels . There is a strong correlation between OSC and fibroblastic factor -23 (FBF-23). Many recent studies have correlated FBF-23 as well as vitamin D levels with some of the pathological conditions such as chronic kidney failure, atherosclerosis, and diabetes. They stated possible interrelationships between insulin resistance, Hyperinsulinemia, and/or lower VD3 levels may lead to decreased serum FGF-23 concentrations in obese children and adolescents. Therefore, serum FGF-23 has been suggested to be a potential indicator of subclinical atherosclerosis in patients with gestational diabetes mellitus. Based on these data, we expect that a high dose of vitamin D will significantly influence the association between A1c with FGF-23 levels in people with vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included males and females in the age range of 22-55 years with a medical diagnosis of vitamin D deficiency.

Exclusion Criteria:

* subjects with any chronic disease such as kidney failure, CVD, diabetes, blood disorders, or immune problems, including autoimmune diseases, chronic or severe infections will be excluded.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
FGF-23 | 10 weeks
  plasma levels
A1c | 10 weeks
  plasma percentage

SECONDARY OUTCOMES:
Osteocalcin | 10 weeks
  plasma levels
25OHD | 10 weeks
  serum

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Study Chair — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan; Sara Al-imam, MSc, Principal Investigator — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan
Locations (1):
- Mahmoud S Abu-Samak, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abu-Samak MS, AbuRuz ME, Masa'Deh R, Khuzai R, Jarrah S. Correlation of selected stress associated factors with vitamin D deficiency in Jordanian men and women. Int J Gen Med. 2019 Jun 28;12:225-233. doi: 10.2147/IJGM.S198175. eCollection 2019. PMID 31303782
- [Result] Al-Shaer AH, Abu-Samak MS, Hasoun LZ, Mohammad BA, Basheti IA. Assessing the effect of omega-3 fatty acid combined with vitamin D3 versus vitamin D3 alone on estradiol levels: a randomized, placebo-controlled trial in females with vitamin D deficiency. Clin Pharmacol. 2019 Feb 4;11:25-37. doi: 10.2147/CPAA.S182927. eCollection 2019. PMID 30787641
- [Result] Abu-Hasheesh MO, Abu-Samak MS, Al-Matubsi HY, Jaradeh MS, Jarrah SS, Khuzaie RF. Association of parental history of type 2 diabetes mellitus with leptin levels in Jordanian male youths. Saudi Med J. 2010 Aug;31(8):882-6. PMID 20714685
- [Result] Abu-Taha M, Dagash R, Mohammad BA, Basheiti I, Abu-Samak MS. Combined Effect Of Coffee Consumption And Cigarette Smoking On Serum Levels Of Vitamin B12, Folic Acid, And Lipid Profile In Young Male: A Cross-Sectional Study. Int J Gen Med. 2019 Nov 22;12:421-432. doi: 10.2147/IJGM.S213737. eCollection 2019. PMID 31819593